CLINICAL TRIAL: NCT01405807
Title: Alemtuzumab for ANCA Associated Refractory Vasculitis - a Study of Safety and Efficacy
Brief Title: Alemtuzumab for ANCA Associated Refractory Vasculitis
Acronym: ALEVIATE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Dr David Jayne, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AL1.1; 2009-017087-17 (EudraCT Number)
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Vasculitis; Microscopic Polyangiitis; Granulomatosis With Polyangiitis; Wegener's
Keywords: Vasculitis; ANCA; Refractory
MeSH Terms: conditions — Vasculitis; Microscopic Polyangiitis; Granulomatosis with Polyangiitis | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alemtuzumab - high dose (60mg) (Experimental): Alemtuzumab 30mg will be administered on Day 1 and Day 2 at 0 and 6 months
  Interventions: Drug: Alemtuzumab
- Alemtuzumab - low dose (30mg) (Experimental): Alemtuzumab 15mg will be administered on Day 1 and Day 2 at 0 and 6 months
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab will be administered on Day 1 and Day 2 at 0 and 6 months
  Other Names: Campath 1H

SUMMARY:
Overview:

This open label, randomized, multi-centre study will enroll and treat 24 patients with refractory AAV.

Aims:

To determine the clinical response and severe adverse event rates associated with alemtuzumab therapy among patients with relapsing or refractory ANCA associated vasculitis (AAV).

Hypothesis:

Treatment with alemtuzumab induces sustained remission in AAV and will reduce immunosuppressive and steroid exposure.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of AAV, according to a standardized definition
2. Active vasculitis with at least one severe or three non severe items of BVAS/WG activity (equivalent to BVAS/WG>3)
3. Previous therapy with either cyclophosphamide or methotrexate, in combination with prednisolone for at least 3 months.

Exclusion Criteria:

1. Age less than 18 or greater than 60 years
2. Creatinine > 150μmol/l (1.7mg/dl)
3. Total white count < 4x109/l or lymphocyte count < 0.5x109/l, or IgG < 5g/L, or neutrophil count < 1.5x109/l.
4. Severe lung haemorrhage with hypoxia (<85% on room air)
5. Severe gastrointestinal, central nervous system or cardiac vasculitis
6. Previous therapy with:

   1. Alemtuzumab at any time
   2. IVIg, infliximab, etanercept, adalimumab, abatacept, anti-thymocyte globulin or plasma exchange in past three months
   3. Rituximab within the past 6 months
7. Intensive care unit requirement
8. Active infection with HIV, hepatitis B or hepatitis C or other infection requiring parenteral or long-term oral antibiotics
9. History of ITP or platelet count at screening below 50,000 x 106/l
10. Pregnancy or inadequate contraception in pre-menopausal women
11. Breast feeding
12. Any condition judged by the investigator that would cause the study to be detrimental to the patient.
13. Any other multisystem autoimmune disease including Churg Strauss angiitis, systemic lupus erythematosus, anti-GBM disease and cryoglobulinaemia
14. Any previous or current history of malignancy (other than resected basal cell carcinoma)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a vasculitis response at 6 months | 6 months
  Response includes patients in complete and partial remission. Complete remission (CR) is defined as a BVAS/WG of 0 for at least one month. Partial response (PR) is the absence of severe BVAS/WG items and at least 50% fall in BVAS/WG score from baseline.
Proportion of patients with a severe adverse event | 6 months

SECONDARY OUTCOMES:
Proportion of patients with treatment failure | 12 months
  Treatment failure is defined as the failure to achieve a vasculitis response by six months or a vasculitis relapse between 6 and 12 months
Combined damage assessment (CDA) scores | 12 months
Non severe adverse events | 12 months
Cumulative dose of corticosteroids | 12 months
Time to remission | 6 months
  Complete and partial
Relapse | 12 months
Change in SF-36 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David RW Jayne, MD MRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, University of Cambridge NHS Foundation Trust, Cambridge, United Kingdom

REFERENCES:
- [Derived] Gopaluni S, Smith R, Goymer D, Cahill H, Broadhurst E, Wallin E, McClure M, Chaudhry A, Jayne D. Alemtuzumab for refractory primary systemic vasculitis-a randomised controlled dose ranging clinical trial of efficacy and safety (ALEVIATE). Arthritis Res Ther. 2022 Apr 1;24(1):81. doi: 10.1186/s13075-022-02761-6. PMID 35365179